CLINICAL TRIAL: NCT02617160
Title: Evaluation of Automated Insulin Pump Settings Using the Advisor Pro (Previously Called) MD-Logic Pump Advisor-three Segments Study
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The required data was obtained and there was no need to collect further data
Sponsor: Rabin Medical Center (Other)
Collaborators: Novo Nordisk A/S (Industry); DreaMed (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RMC059315ctil
Record Dates: First submitted 2015-11-23; First posted 2015-11-30 (Estimated); Last update posted 2018-12-21 (Actual); Status verified 2018-12

CONDITIONS: Type 1 Diabetes
Keywords: Insulin Pump Treatment; Type 1 Diabetes; Insulin Pump Setting; Pump Advisor
MeSH Terms: conditions — Diabetes Mellitus, Type 1 | interventions — Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- MD Logic Pump Advisor (Experimental): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the MD-Logic Pump Advisor
  Interventions: Device: MD-Logic Pump Advisor
- Control Group-Medical guided recommendations (Active Comparator): Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted by the medical team in accordance to the regular practice
  Interventions: Other: Control Group

INTERVENTIONS:
Device: MD-Logic Pump Advisor — Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted using the MD-Logic Pump Advisor
  Arms: MD Logic Pump Advisor
Other: Control Group — Insulin pump settings (i.e, basal plan, correction factor, carbohydrate ratio and insulin activity time) will be adjusted by the medical team in accordance to the regular practice
  Arms: Control Group-Medical guided recommendations

SUMMARY:
Pump therapy is gaining popularity as a treatment mode for patients with type 1 diabetes. Utilizing pump therapy requires the development and application of a new spectrum of theoretical knowledge and practical skills by the patient. Furthermore, occasionally there is a need to tailor the pump settings, i.e. the insulin correction factor, carbohydrate ratio, basal plan and insulin activity time, in order to optimize and improve glucose control. These adjustments are based on collected information including insulin delivery, blood glucose measurements, continuous glucose monitoring data, meals and so on. Analyzing this multitude of information and data is overwhelming for many of the patients, caregivers and health care providers. Unfortunately, not all physicians have the needed expertise to fully fulfill this task, and for those who do, it is time consuming. Thus, a summary of the data with insulin dose adjustment suggestions is missing. An automated tool for pump setting adjustments will improve glycemic control without escalating the burden on patients and the health care system. Such advisor can assist the professional team during routine follow-up and the patients between visits.

To address this challenge, the investigators developed the MD-Logic Pump Advisor (MDPA), which automatically analyses treatment information, learns patient's needs and accordingly suggests adjustments in insulin dosing. The MDPA uses information gathered from glucose monitoring, insulin dosing and meal data during daily routine home care. Following a 5 minute data collection and analysis, the algorithm learns and suggests pump-setting changes for optimization of glucose control.

This study aims to evaluate the efficacy and safety of the Advisor Pro. The study will include three segments:

Segment A - a randomized controlled parallel study, Segment B- a clinic prospective study during which the Advisor Pro will be evaluated during routine clinical visits as an added tool for physicians and Segment C- a clinical prospective parallel study for patients treated with pump therapy and SMBG only.

ELIGIBILITY:
Inclusion Criteria:

* Documented Type 1 Diabetes for at least 1 year prior to study enrollment
* Segment A:Subjects aged ≥ 10 years and up to 25 years Segment B: Subjects aged ≥ 6 years Segment C: Subjects aged ≥ 6 years and up to 30 years
* HbA1c at inclusion ≤ 11%
* Insulin pump therapy for at least 4 months for segment A and C and at least 3 months for segment B
* BMI Standard Deviation Score - below the 97th percentile for age
* Subjects have continuous glucose monitoring data for at least 2-3 weeks before the clinic regular visit (for segment B only)
* Without routine sensor use (for segment C only)
* Subjects willing to follow study instructions

Exclusion Criteria:

* An episode of diabetic keto-acidosis within the month prior to study entry
* Severe hypoglycemia resulting in seizure or loss of consciousness in the month prior to enrollment
* Concomitant diseases/ treatment that influence metabolic control
* Significant diseases /conditions including psychiatric disorders and substance abuse that in the opinion of the investigator is likely to affect the subjects ability to complete the study or compromise patients safety
* Participation in any other interventional study
* Known or suspected allergy to trial products
* Female subject who is pregnant or planning to become pregnant within the planned study duration.

Ages: 6 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Actual)
Dates: Start 2016-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Percentage of glucose readings within range of 70-180 mg/dl | Day 90 for segments A and C and day 30 for segment B

SECONDARY OUTCOMES:
Percentage of glucose readings below 60 mg/dl | Day 90 (for segments A and C only)
HbA1c levels | Day 90 (for segments A and C only)
Percentage of glucose readings below 54 mg/dl | Day 30 for segment B and Day 90 for segment C
Percentage of glucose readings below 50 mg/dl | Day 30 (for segment B only)

OTHER OUTCOMES:
The percentage of glucose readings below 70 mg/dl | Day 90 for segments A and C and Day 30 for segment B
The percentage of glucose readings above 240 mg/dl | Day 90 for segments A and C and day 30 for segment B
The percentage of glucose readings above 180 | Day 90 for segments A and C and day 30 for segment B
Number of unexplained hyperglycemic events | Day 90 (segments A and C only)
Area above the curve of 180 mg/dl | Day 90 (Segments A and C only)
Area under the curve of 70 mg/dl | Day 90 (segments A and C only)
Mean sensor blood glucose | Day 90 for segments A and C and day 30 for segment B
Glucose variability measured by Standard Deviation (SD) | Day 90 for segments A and C and day 30 for segment B
Number of recommendations for changes in settings per patient and per iteration | Day 90 for segments A and C and day 30 for segment B
Number of physician override advisor recommendations | Day 90 for segments A and C and day 30 for segment B
  Number of physician override advisor recommendations only for the intervention arm during each iteration and for all insulin dose changes
Time duration needed for the physician to give his recommendations | Day 90 (segments A and C only)
Quality of Life Score in QoL Questionnaire | Day 90 (segment A only)
Diabetes Treatment Satisfaction Score in Diabetes Treatment Satisfaction Questionnaire (DTSQ) | Day 90 ( segment A only)
Device Satisfaction | Day 30 ( Segment B only)
  Device Satisfaction evaluated by the Healthcare Professional Survey

CONTACTS AND LOCATIONS:
Overall Officials: Moshe Phillip, MD, Prof, Principal Investigator — Rabin Medical Center
Locations (1):
- Schneider Medical Center, Petah Tikva, Israel